CLINICAL TRIAL: NCT01404351
Title: A Prospective, Randomized, Controlled Superiority Study to Evaluate Use of the PEAK PlasmaBlade® 4.0 in Bilateral Breast Reduction
Brief Title: Use of the PEAK PlasmaBlade 4.0 in Bilateral Breast Reduction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to the acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-00133
Record Dates: First submitted 2011-07-25; First posted 2011-07-28 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Macromastia (Symptomatic)
Keywords: Reduction mammaplasty; Breast reduction; PlasmaBlade; PEAK
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEAK PlasmaBlade (Experimental)
  Interventions: Device: PEAK PlasmaBlade
- Standard of Care (Active Comparator): The Standard of Care arm will consist of the scalpel for the skin incision and traditional electrosurgery for subcutaneous dissection.
  Interventions: Procedure: Scalpel and Traditional Electrosurgery

INTERVENTIONS:
Device: PEAK PlasmaBlade
  Arms: PEAK PlasmaBlade
Procedure: Scalpel and Traditional Electrosurgery
  Arms: Standard of Care

SUMMARY:
The objective of this clinical study is to evaluate the operative performance of the PEAK PlasmaBlade® 4.0 during bilateral breast reduction; to monitor and record post-operative pain, adverse events and skin scarring following surgery; and to compare these outcomes to the HARMONIC SYNERGY® BLADE.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70
2. Physically healthy, stable weight
3. No smoking <1 month prior to surgery and during study.
4. Desiring bilateral breast reduction
5. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
6. Subject must be willing and able to comply with specified follow-up evaluations.
7. Female subjects must either be incapable of reproduction, or taking acceptable measures to prevent pregnancy and have a negative pregnancy test prior to participation in the study.

Exclusion Criteria:

1. Age younger than 18 or greater than 70 years old
2. Anticoagulation therapy which cannot be discontinued
3. Smoking <1 month prior to surgery or during study
4. Infection (local or systemic)
5. Cognitive impairment or mental illness
6. Severe cardiopulmonary deficiencies
7. Known coagulopathy
8. Immunocompromised
9. Prior history of breast cancer
10. Kidney disease (any type)
11. Currently taking any medication known to affect healing
12. Subjects who are status-post gastric banding or gastric bypass
13. Currently enrolled in another investigational device or drug trial
14. Unable to follow instructions or complete follow-up

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference in pain | 24 hours and first 10 days post-op
  The primary endpoint will be the difference in pain between the Harmonic and PlasmaBlade operative sites. The primary efficacy variable will be pain at each treatment arm operative site, as measured by visual analog scale for 24 hours post-operatively and for 10 post-op days twice daily.

SECONDARY OUTCOMES:
Operative performance | Intraoperatively on day 0
  Dissection time (normalized), estimated blood loss, use of traditional device for bleeding control, volume of tissue resection.
Adverse events | 1 month post-operatively
  Monitoring for adverse events following surgery, including hematoma, seroma, wound dehiscence, etc.
Cutaneous scarring | Up to one year post-operatively
  Scar width, quality, pigmentation, elevation, nodularity, thickness, and cosmetic appearance will be blindly evaluated by subject and independent observers.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Gonyon, MD, Principal Investigator — Gonyon Cosmetic & Plastic Surgery, PC
Locations (1):
- Gonyon Cosmetic & Plastic Surgery, PC, Johnstown, Colorado, United States